CLINICAL TRIAL: NCT05394155
Title: Determination of Leucine Requirement in Young Men and Women Using the Indicator Amino Acid Oxidation (IAAO) Method
Brief Title: Leucine Requirement in Adult Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Associate Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000078896
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: Leucine; amino acid; nutrition; requirement
MeSH Terms: interventions — Leucine

STUDY DESIGN:
Intervention Model Description: Repeated measures study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leucine intake (Experimental): For this study, each participant will be randomly assigned to receive up to 7 intake levels of leucine, ranging from 10 to 75 mg/kg/d.
  Interventions: Dietary Supplement: Leucine

INTERVENTIONS:
Dietary Supplement: Leucine — 7 intake levels of leucine, ranging from 10 to 75 mg/kg/d.

SUMMARY:
The purpose of the study is to determine the body's nutritional need for the essential amino acid, leucine, in adult men and women 18 to 39 years of age.

DETAILED DESCRIPTION:
The experimental design will be based on the minimally invasive IAAO model (12). Each participant will be studied at a minimum of 4 and up to 7, randomly assigned, intake levels of leucine.

Subjects will be weighed at the pre-study assessment and at the start of each IAAO study day to ensure accurate prescription of diets and isotopes, and to confirm weight maintenance throughout the study.

Each study will consist of a 2-day adaptation period to a prescribed diet in accordance with the energy requirement of the subject and 1-study day. The diet will provide an adequate amount of protein, of 1 g protein∙kg-1∙d-1. The 2-day adaptation period is to allow the body to adapt to an adequate amount of protein as it has been shown that protein kinetics is altered without it. Following the 2 days of adaptation is the study day where leucine intake will be randomly assigned and phenylalanine (Phe) kinetics will be measured with the use of L-[1-13C]phenylalanine. On this day, VCO2 will be measured by calorimetry immediately after the 5th meal for a period of 20 minutes, and a 15ml blood sample will be collected at the end of each study visit to measure plasma amino acid levels, insulin, and glucose in males and females and progesterone, and estrogen in females.

For female participants, each level of intake will be studied both in the luteal and follicular phase of their menstrual cycle (up to 14 studies in total). For the follicular phase, the study will be conducted 3-7 days immediately after the 1st day of menstrual bleeding. For the luteal phase, the study will be conducted 4-7 days before the onset of next menstrual bleeding. The IAAO study day of the luteal phase will be set on the basis of each subject's length of their menstrual cycle, and the length and regularity of their cycle will be determined during the pre-study assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males, 18 to 39 years of age.
2. Healthy adult females, 18 to 39 years of age with regular menstrual cycles within in the last 12 months.
3. Willingness to participate in the study and completed the screening procedures (height, weight, fasting blood sample and medical history questionnaire).
4. No recent history of weight loss
5. BMI between 18.5 - 27 kg/m 2
6. Absence of chronic disease or acute illness that could affect protein and AA metabolism (diabetes, cancer, liver or kidney disease, HIV, acute cold or flu, COVID-19, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications).
7. Non-smoking
8. Willingness to consume the diet provided.

Exclusion Criteria:

1. Presence of disease known to affect protein and AA metabolism (diabetes, cancer, liver or kidney disease, HIV, acute cold or flu, Covid-19, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications).
2. On medications known to affect protein and amino acid metabolism (steroids) or taking oral contraceptive pills or other birth control devices that would affect sex hormone profiles over the last 2 years.
3. Pregnant or lactating women.
4. Recent significant weight loss; ≥ 5% of body with in the last 3 months.
5. Individuals on weight reducing diets.
6. Inability to tolerate the diet
7. Unwilling to have blood drawn from a venous access, or using a ventilated hood indirect calorimeter for the purposes of the study.
8. Significant coffee consumption of more than 2 cups/day
9. Significant alcohol consumption of more than one drink/day
10. Failure to disclose any of the information needed to assess eligibility.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
F13CO2 | 4.5 hours during study visits
  Rate of appearance of labelled carbon dioxide (13CO2) in breath from the oxidation of 13C-Phenylalanine

SECONDARY OUTCOMES:
13C-phenylalanine enrichment | 4.5 hours during study visits
  urinary 13C-phenylalanine enrichment
Plasma amino acid concentrations | at end of each study visit
  To assess the effect of amino amino acid intake on plasma amino acid concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, PhD, RD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szwiega S, Pencharz PB, Xu L, Kong D, Tomlinson C, Elango R, Courtney-Martin G. Leucine requirement determined in healthy young adult males using the indicator amino acid oxidation method. Am J Clin Nutr. 2024 Nov;120(5):1063-1070. doi: 10.1016/j.ajcnut.2024.08.022. Epub 2024 Aug 28. PMID 39209155